CLINICAL TRIAL: NCT05838924
Title: Changing Lower Back Pain Through Virtual Reality: a Randomised Clinical Controlled Trial
Brief Title: Changing Lower Back Pain Through Virtual Reality
Acronym: CLEVER-BODY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-63
Record Dates: First submitted 2023-04-03; First posted 2023-05-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: Virtual Reality; Physical Activity; Range of movement; Pain; Disability; Kinesophobia
MeSH Terms: conditions — Low Back Pain; Motor Activity; Pain; Kinesiophobia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity + Virtual Reality (Experimental): A program of 8 VR exercises will be applied, of a therapeutic nature, based on the applied exercises of the "Back School", aimed at gaining strength, stability, mobility and flexibility of the abdomino-lumbo-pelvic region and the lower extremities. For each exercise, the VR goggles will manipulate the visual proprioceptive information by modifying the perceived degree of lumbar flexion and extension, i.e., in the VR goggles they will perceive that your movements are different from what you are actually doing.
  Interventions: Other: PHYSICAL ACTIVITY + VIRTUAL REALITY
- Physical Activity (Active Comparator): The same therapeutic exercise program will be applied as the experimental group, but without VR. The training methodology and progression of loads, evaluations and supervision by the physiotherapist will also be the same.
  Interventions: Other: PHYSICAL ACTIVITY

INTERVENTIONS:
Other: PHYSICAL ACTIVITY + VIRTUAL REALITY — The VR therapeutic exercise program will be implemented for 6 weeks at a frequency of 2 sessions per week with the aim of improving pain and disability, kinesiophobia, range of motion (ROM), catastrophizing, quality of life, and physical fitness. This group will perform the 8 VR exercises of "Back School" by manipulating visual proprioceptive information during all lumbar movements. They will be performed in 2 sets whose intensity and repetitions will be configured and individualized by a self-reported rating of perceived exertion (RPE) through the Borg 6-20 scale. The appropriate training intensity is established with an RPE score between 13 and 17; for this reason, the first 2 weeks will work at an RPE of 14, the 3rd and 4th weeks at an RPE of 15; and finally, the last 2 weeks will work at an RPE of 16. The first 3 weeks will work without additional load, and the last 3 weeks will work with weights, increasing their weekly load individually.
  Arms: Physical Activity + Virtual Reality
Other: PHYSICAL ACTIVITY — The 8 therapeutic exercise program will be implemented for 6 weeks at a frequency of 2 sessions per week with the aim of improving pain and disability, kinesiophobia, range of motion (ROM), catastrophizing, quality of life, and physical fitness. This group will perform the 8 exercises of "Back School" without VR. They will be performed in 2 sets whose intensity and repetitions will be configured and individualized by a self-reported rating of perceived exertion (RPE) through the Borg 6-20 scale. The appropriate training intensity is established with an RPE score between 13 and 17; for this reason, the first 2 weeks will work at an RPE of 14, the 3rd and 4th weeks at an RPE of 15; and finally, the last 2 weeks will work at an RPE of 16. The first 3 weeks will work without additional load, and the last 3 weeks will work with weights, increasing their weekly load individually.
  Arms: Physical Activity

SUMMARY:
The main objective of this randomized controlled trial is to investigate the efficacy of a 6-week therapeutic exercise program, performed with virtual reality (VR) manipulating visual proprioceptive information during all lumbar movements in the different therapeutic exercises (experimental group), on pain and disability, kinesiophobia, range of motion (ROM), catastrophizing, quality of life, and physical fitness in patients with chronic non-specific low back pain compared to the same therapeutic exercise program without VR (control group).

DETAILED DESCRIPTION:
Chronic pain is considered an urgent global public health problem. One of the most prevalent chronic pain pathologies worldwide is low back pain (LBP). Kinesophobia (fear of movement) has been largely associated with pain intensity, disability, worse quality of life and chronification in LBP; while physical reconditioning has been proposed in clinical practice as a key element in the treatment of LBP.(20-22) However, the efficacy of physical reconditioning programs developed so far would require considerable improvement. The induction of illusions in virtual reality (VR) through visual cues could be a valid alternative to evoke motion illusions and be able to modify proprioceptive integration, acting on kinesiophobia, in turn. The main objective of this randomized controlled trial is to investigate the efficacy of a 6-week therapeutic exercise program, performed with VR manipulating visual proprioceptive information during all lumbar movements in the different therapeutic exercises (experimental group), on pain and disability, kinesiophobia, range of motion (ROM), catastrophizing, quality of life, and physical fitness in patients with chronic non-specific low back pain compared to the same therapeutic exercise program without VR (control group).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic non-specific lower back pain according to the European COST B13 guideline.
* Pain score of 3 or higher on the Numeric Rating Scale (NRS) in the last 6 months.

Exclusion Criteria:

* Presence of spinal tumor.
* Presence of infection.
* Presence of fracture.
* Presence of systemic disease.
* Presence of fibromyalgia.
* Presence of cauda equina syndrome.
* Previous spinal surgery.
* Presence of musculoskeletal injuries of the lower extremities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Low back pain | At six weeks
  Measured with a Visual Analogue Scale (0-10 points). Higher scores mean a worse pain.
Range of movement | At six weeks
  Measured with an electrogoniometer
Disability | At six weeks
  Measured with the Roland Morris Questionnaire (0-24 points). Higher scores mean a worse disability.

SECONDARY OUTCOMES:
Physical activity | At six weeks
  Measured with the International Physical Activity Questionnaire (short-form). This is a 7-item scale used to assess physical activity. Results are divided into different activity levels (low or inactive, moderate, and high activity), and scores are obtained by multiplying the duration of physical activity by the intensity of a task that is metabolically equivalent for each activity level in the last 7 days.
The Quality of life | At six weeks
  Measured with the Euro Quality of life five dimensions with five levels questionnaire (-0.59 to 1.0). Higher scores mean a better quality of life.
Kinesophobia | At six weeks
  Measured with the Fear Avoidance Beliefs Questionnaire
Catastrophizing | At six weeks
  Measured with the Pain Catastrophizing Scale (0-52 points). Higher scores indicate higher levels of fear-avoidance beliefs.
Physical capacity | At six weeks
  Measured with the Sit-to-Stand 60 test. The STS-60 measures the number of times an individual can sit and stand up from a chair in 60 seconds. Higher number of repetitions indicate higher physical capacity.

CONTACTS AND LOCATIONS:
Overall Officials: JUAN JOSÉ AMER-CUENCA, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harvie DS, Broecker M, Smith RT, Meulders A, Madden VJ, Moseley GL. Bogus visual feedback alters onset of movement-evoked pain in people with neck pain. Psychol Sci. 2015 Apr;26(4):385-92. doi: 10.1177/0956797614563339. Epub 2015 Feb 17. PMID 25691362